CLINICAL TRIAL: NCT03659370
Title: Chinese Herbal Fumigation in Conjunction With Acupuncture for the Knee Osteoarthritis: a Three-armed Randomized Controlled Trial
Brief Title: Chinese Herbal Fumigation With Acupuncture for the Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fumigation 2016
Record Dates: First submitted 2018-08-20; First posted 2018-09-06 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee; Fumigation; Acupuncture
MeSH Terms: conditions — Osteoarthritis | interventions — Fumigation; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fumigation Full (Active Comparator): Full Fumigation after acupuncture, 2 times per week, for 4 weeks.
  Interventions: Other: Fumigation
- Fumigation 1/16 (Active Comparator): 1/16 Fumigation after acupuncture, 2 times per week, for 4 weeks.
  Interventions: Other: Fumigation
- Acupuncture (Active Comparator): Acupuncture only, 2 times per week, for 4 weeks.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Fumigation — use Fumigation to increase the improvement of osteoarthritis of knee
  Arms: Fumigation 1/16; Fumigation Full
Other: Acupuncture — Acupuncture
  Arms: Acupuncture

SUMMARY:
To evaluate the effect of fumigation in conjunction with acupuncture for knee osteoarthritis, participators were collected from acupuncture and Chinese traumatology clinic at Linsen Chinese Medicine and Kunming Branch, Taipei City Hospital. Participators were randomized into 3 groups, one for acupuncture with fumigation, one for acupuncture with diluted fumigation, one for acupuncture only.

DETAILED DESCRIPTION:
Patient population. Between June 2015 and November 2017, research subjects were recruited via poster display and clinician referral, to participate in a three-armed, randomized, controlled trial to be conducted in the Traumatology Department Linsen Chinese Medicine and Kunming Branch, Taipei City Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of knee diagnosed by X-ray films
* According Ahlbäck System, more than stage1
* The Visual Analogue Scale of pain over 20mm in 100mm

Exclusion Criteria:

* The Visual Analogue Scale of pain less than 20mm in 100mm
* Received injection or scope treatment over knees
* Received more than 3 times of operation
* With severe inflammation (including fever, fluid, pus, gout, Rheumatic arthritis, etc.)
* With sever systemic diseases (including metastatic cancer, coronary artery disease, lung disease, etc.)
* With history of skin problem after other thermal treatment
* Under other experiments
* Women with pregnant, breastfeeding or prepare for pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale of pain | This numeric measure is assed and recorded pre and post intervention at each of the study protocols bi-weekly interventions over (4) weeks, for a maximum of (8) sessions and a total of (16) measurements per individual patient.
  This scale is used to asses change in pain intensity between pre and post intervention measures and change against established baseline measures. Patients are asked to rate their pain by choosing a number along a horizontal line of fixed length (100mm). The number scale ranges from 0-10, with 0 representing 'no pain' and 10 being 'worst pain possible'.

SECONDARY OUTCOMES:
Questionnaire | This questionnaire is administered and recorded after patients have been enrolled in the trial and prior to their first intervention to establish a baseline. At the completion of the protocol's full course of treatment, bi-weekly treatment over (4) weeks
  Record Questionnaire before the study starting and after study finished

CONTACTS AND LOCATIONS:
Overall Officials: CHUNG-HUA HSU, PhD, Study Chair — Taipei City Hospital, Linsen Chinese Medicine & Kunming Branch,
Locations (1):
- Linsen Chinese Medicine and Kunming Branch, Taipei City Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No